CLINICAL TRIAL: NCT05039632
Title: Phase I/II Randomized Study of NBTXR3 Activated by Abscopal or RadScopal Radiation in Combination With Immunotherapy (Anti-PD-1/L-1) for Patients With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0618; NCI-2021-09077 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0618 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-02; First posted 2021-09-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Neoplasm in the Liver; Metastatic Malignant Neoplasm in the Lung; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (NBTXR3, Abscopal, Anti PD-1 / PD-L1 (Experimental): COHORT I: Patients receive NBTXR3 intratumorally on day 1. Patients also receive ( anti-PD-1/L-1) intravenously (IV) on day 8. Beginning day 15, patients undergo Abscopal radiation therapy over 1-2 weeks. Cycles with ( anti-PD-1/L-1) repeat every 3-6 weeks per standard of care up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Hafnium Oxide-containing Nanoparticles NBTXR3; Radiation: Radiation Therapy
- Cohort II (NBTXR3, RadScopal, Anti PD-1 / PD-L1 (Experimental): COHORT II: Patients receive NBTXR3 intratumorally on day 1. Patients also receive ( anti-PD-1/L-1) IV on day 8. Beginning day 15, patients undergo RadScopal radiation therapy over 1-2 weeks. Cycles with ( anti-PD-1/L-1)repeat every 3-6 weeks per standard of care up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Hafnium Oxide-containing Nanoparticles NBTXR3; Radiation: Radiation Therapy

INTERVENTIONS:
Other: Hafnium Oxide-containing Nanoparticles NBTXR3 — Given intratumorally
  Other Names: NBTXR3
Radiation: Radiation Therapy — Undergo Abscopal radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Cohort I (NBTXR3, Abscopal, Anti PD-1 / PD-L1
Radiation: Radiation Therapy — Undergo RadScopal radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Cohort II (NBTXR3, RadScopal, Anti PD-1 / PD-L1

SUMMARY:
This phase I/II trial studies the side effects and possible benefits of NBTXR3, radiation therapy, Anti PD-1 / PD-L1 in treating patients with solid tumor that has spread to the lung (lung metastases) and/or liver (liver metastases). NBTXR3 may help make tumor cells more sensitive to the radiation therapy. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Immunotherapy with Anti PD-1 / PD-L1 monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving NBTXR3, radiation therapy, Anti PD-1 / PD-L1 may help to control the disease.

DETAILED DESCRIPTION:
Primary Objective

Phase I & II

• To evaluate efficacy and safety of NBTXR3 activated by radiation (Abscopal or RadScopal™) in combination with immunotherapy ( anti-PD-1/L-1)

Secondary Objective:

* To evaluate the safety profile of NBTXR3 activated by radiation (Abscopal or RadScopal™) in combination with immunotherapy ( anti-PD-1/L-1).
* To evaluate time-to-event outcomes of NBTXR3 activated by radiation (Abscopal or RadScopal™) in combination with immunotherapy ( anti-PD-1/L-1).

Exploratory Objectives:

I. To evaluate radiomic measurements with outcomes of study treatments.

II. To evaluate biomarkers of response in subjects after receiving study treatment.

OUTLINE: Patients are randomized to 1 of 2 cohorts.

COHORT I: Patients receive NBTXR3 intratumorally on day 1. Patients also receive ( anti-PD-1/L-1) intravenously (IV) on day 8. Beginning day 15, patients undergo Abscopal radiation therapy over 1-2 weeks. Cycles with ( anti-PD-1/L-1) repeat every 3-6 weeks per standard of care up to 2 years in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive NBTXR3 intratumorally on day 1. Patients also receive ( anti-PD-1/L-1) IV on day 8. Beginning day 15, patients undergo RadScopal radiation therapy over 1-2 weeks. Cycles with ( anti-PD-1/L-1)repeat every 3-6 weeks per standard of care up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for up to 2 years post-radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic disease in the lung and/or liver, or soft tissue from any primary malignancy considered incurable by local therapies.

   a. One prior anti-PD-1/L1 therapy allowed.
2. The target lesion(s) must be measurable as per irRECIST and repeated measurements at the same anatomical location should be achievable.

   a. Participant must have at least 2 measurable lesions at screening. i. Abscopal cohort: At least one lesion will receive NBTXR3 and high dose radiation (high dose target lesion). The other lesion(s) (non-treated target lesion) will be followed for response and it will not receive NBTXR3 or RT.

   ii. RadScopal™ cohort: At least one lesion will receive NBTXR3 and high dose radiation (high dose target lesion). The other lesion(s) will only receive low dose radiation (low dose target lesion).
3. Amenable to undergo the image guided (EBUS or CT or MRI) intratumoral injection of NBTXR3, in up to two (2) high dose target lesions, as determined by the investigator or treating physician at screening.

   a. Intratumoral NBTXR3 injections only allowed in lung or liver lesions.
4. Selected high and low dose target lesions must be amenable to receive radiation therapy as determined by the investigator or treating radiation oncologist.

   1. Allowed high dose RT regimens are 50 Gy in 4 fractions or 60 Gy in 10 fractions
   2. Allowed low dose RT for RadScopal™ cohort is 1.4 Gy per fraction for 4 - 5 fractions to only low dose-target lesion(s) determined by the investigator or treating physician.
5. Patients can receive radiation therapy for symptomatic metastatic disease prior to enrollment or during the study a.
6. Age ≥ 18 years
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
8. Laboratory Values at screening:

   1. Hemoglobin ≥ 9.0 g/dL
   2. Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
   3. Platelet count ≥ 100,000/mm3
   4. Leukocytes ≥ 1500/mm3
   5. Creatinine ≤ 1.5 x upper limit of normal (ULN)
   6. Calc. creatinine clearance > 30mL/min
   7. Total bilirubin ≤ 2.0 mg/dL
   8. AST / ALT ≤ 2.0 x upper limit of normal (ULN) or ≤ 3 x ULN for patients with liver metastases
9. For participants to be treated for lung metastases, adequate lung function with expiratory volume in 1 second (FEV1) ≥ 0.8L or ≥ 35% predicted and carbon monoxide diffusing capability (DLCO) ≥ 40% with or without bronchodilator within 30 days prior to NBTXR3 injection. Participants to be treated for liver metastasis a pulmonary function test is not required.
10. Patients who meet the criterion above without oxygen (02), but need acute (started within 7 ± 3 days) supplemental oxygen due to tumor-caused obstruction/hypoxia are eligible, provided the amount of the O2 needed has been stable.
11. Negative urine or serum pregnancy test ≤ 7 days prior to NBTXR3 injection in all women of child-bearing potential (WOCBP). WOCBP must agree to follow instructions for method(s) of contraception for the duration the entire study period and 160 days (~5.33 months) after the last dose of anti-PD-1/L-1 treatment. Local laws and regulations may require use of alternative and/or additional contraception methods. WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements but should still undergo pregnancy testing.
12. Signed informed consent form (ICF) indicating that participant understands the purpose of, and procedures required for, the study and is willing to participate in the study.

4.2 Exclusion criteria:

1. Prior radiation therapy received to the selected high dose target lesion(s)

   a. Previous radiation to low dose target lesions allowed as per investigator or treating radiation oncologist discretion.
2. Symptomatic central nervous system metastases and/or carcinomatous meningitis

   a. Participants with previously treated brain metastases may participate if those lesions are radiologically stable (i.e., without evidence of progression for at least 4 weeks by repeat imaging at screening), clinically stable, and without requirement of steroid treatment for at least 14 days prior to NBTXR3 injection.
3. At screening, past medical history of:

   1. Interstitial lung disease
   2. Unresolved organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia)
   3. Any Grade 4 radiation toxicity
   4. Unresolved, radiation or ICI related

   i. Pneumonitis ii. Bronchopulmonary hemorrhage iii. Abdominal hemorrhage e. Unresolved GI related events i. Diverticulitis ii. Colitis iii. Intra-abdominal abscess iv. GI obstructions v. Abdominal carcinomatosis vi. Any known risk factor for bowel perforation
4. History of severe (Grade ≥ 3) immune-related adverse events observed with previous immunotherapy (anti-PD-1/L1) or known sensitivity (Grade ≥ 3) to any excipients.
5. Has received any approved or investigational anti-neoplastic agent or immunotherapy within 2 weeks prior to NBTXR3 injection.

   1. Except anti-PD-1/L1, which will not require a washout window.
   2. A reduced washout window may be considered for therapies with short half-lives (i.e., kinase inhibitors) after discussion with Nanobiotix and investigator.
6. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).

   a. Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement [≤ 10 mg prednisone] therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
7. Any live-virus vaccine used for prevention of infectious diseases administered within 4 weeks prior to NBTXR3 injection.

   1. Except killed-virus Influenza vaccine
   2. Exception of other vaccines (e.g. pneumonia) is at the discretion of the treating physician after conducting a personalized risk assessment on a case by case basis.
8. Prior allogenic stem cell transplantation or organ allograft.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, renal failure, cardiac arrhythmia, or psychiatric illness that would limit compliance with treatment.
10. Known active, uncontrolled (high viral load) HIV or hepatitis B or hepatitis C infection.
11. Female patients who are pregnant or breastfeeding.
12. Women of child-bearing potential and their male partners who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and up to 160 days (~5.33 months) for female participants, and 7 months for males participants or female partners of male participants that are of child-bearing potential, after the last dose of anti-PD-1/L-1.

    a. Acceptable methods of contraception are those that, alone or in combination, result in a failure rate of < 1% per year when used consistently and correctly.
13. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | Up to 4 weeks post radiation therapy
  Descriptive summary tables will be produced.
Objective response rate | Up to 12 weeks post radiation therapy
  Defined as percentage of patients achieving complete or partial response, per immune-related Response Evaluation Criteria In Solid Tumors (irRECIST). The best overall response will be provided per irRECIST criteria and consideration of all imaging assessment is required.

CONTACTS AND LOCATIONS:
Overall Officials: Saumil Gandhi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org